CLINICAL TRIAL: NCT04028687
Title: Post Market Clinical Follow up Study to Provide Safety, Performance and Clinical Benefits Data of the Taperloc Complete Stems
Brief Title: MDR - PMCF Study for Taperloc Complete Stems
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-39H
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthritis; Hip Disease; Hip Fractures; Hip Injuries; Hip Pain Chronic
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Taperloc Complete Stems: Patients that have been implanted with a Taperloc Complete Stem to repair hip malfunction/disease.
  Interventions: Device: Taperloc Complete Stem

INTERVENTIONS:
Device: Taperloc Complete Stem — Patients that have been implanted with a Taperloc Complete Stem to improve hip malfunction/disease.

SUMMARY:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the Taperloc Complete stems when used for primary or revision total hip arthroplasty (implants) at 1,3,5,7 and 10-year follow-up*. Since Taperloc Complete was introduced to the EU in 2010, all available retrospective data will be collected from each patient and a prospective aspect to the study will be necessary to reach the 10-year time point.

DETAILED DESCRIPTION:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance, and clinical benefits of the Taperloc Complete stems when used for primary or revision total hip arthroplasty (implants) at 1,3,5,7 and 10-year follow-up*. Since Taperloc Complete was introduced to the EU in 2010, all available retrospective data will be collected from each patient and a prospective aspect to the study will be necessary to reach the 10-year time point.

The primary objective is to confirm safety of the study products. This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by analyzing recorded patient-reported clinical outcomes measures (PROMs).

*The most recent available data will be used. If any of the listed time points are not available, data will be used from last available time point and follow-up will move forward at the closest available time point

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older and skeletally mature
* Patient must be willing and able to sign IRB approved informed consent
* Patient must have undergone primary or revision hip arthroplasty with the -Taperloc Complete stem according to a cleared indication, which includes the following:
* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques

Exclusion Criteria:

* Off-label use
* Infection
* Sepsis
* Osteomyelitis
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease
* Patient is known to be pregnant or nursing
* Patient is a prisoner
* Patient is a known alcohol or drug abuser
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of patients implanted with the Taperloc Complete Stems in primary or revision total hip arthroplasty according to the approved indications.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2032-02-12 (Estimated); Study Completion 2032-02-12 (Estimated)

PRIMARY OUTCOMES:
Device Safety assessed through the frequency and incidence of revisions, complications and Adverse Events. | Out to 10 Years
  The primary objective of this study is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications and adverse events. Relation of the events to either implant or instrumentation should be specified.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Harris Hip Score | Out to 10 Years
  The HHS is divided into 4 sub-categories; pain (44 points), function (47 points), range of motion (5 points), and absence of deformity (4 points). Patients select a discrete set of answers which correspond to predefined point allocations based on the category. To obtain a final score, these values are summed.
Device Performance and Benefits evaluated through the Oxford Hip Score | Out to 10 Years
  The OHS is a patient-completed, 12-question evaluation. Each item is scored from 1 to 5, with 1 representing best outcome/least symptoms and 5 representing worst outcome/most symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orthopaedic Institute of Henderson, Henderson, Nevada
  - Texas Health Physicians Group, Plano, Texas
  - Proliance Orthopaedics and Sports Medicine, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No